CLINICAL TRIAL: NCT06989086
Title: FearLess in Neuro-Oncology
Brief Title: FearLess in NeuroOncology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Brain Tumor Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-24-21975; 1R34CA286879 (NIH); HM20031650 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2025-05-13; First posted 2025-05-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Primary Malignant Brain Tumor; Glioblastoma (GBM); Astrocytoma; Oligodendroglioma; Caregiver
Keywords: brain tumor
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Delayed treatment control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fearless Immediate Treatment Arm (Experimental): FearLess is a newly developed, empirically-rooted, manualized psychological intervention consisting of an intake + 8 sessions delivered over a 12-week time period. It consists of weekly individual 60- to 90-minute virtual therapy sessions. FearLess will be delivered immediately following enrollment in this arm.
  Interventions: Behavioral: Fearless in Neuro-Oncology
- FearLess Delayed Control Arm (Other): FearLess is a newly developed, empirically-rooted, manualized psychological intervention consisting of an intake + 8 sessions delivered over a 12-week time period. It consists of weekly individual 60- to 90-minute virtual therapy sessions. In this arm, the FearLess intervention will begin following a 12-week no-treatment period.
  Interventions: Behavioral: Fearless in Neuro-Oncology

INTERVENTIONS:
Behavioral: Fearless in Neuro-Oncology — FearLess is a newly developed, empirically-rooted, manualized psychological intervention consisting of an intake + 8 sessions delivered over a 12-week time period. It consists of weekly individual 60- to 90-minute virtual therapy sessions.

SUMMARY:
The overarching goal of this project is to assess the feasibility, acceptability, and appropriateness of recruitment methods, target population, and a waitlist design to finalize the protocol of FearLess in primary malignant brain tumor patients and caregivers

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility, acceptability, appropriateness (FAA) of recruitment methods, study population, and waitlist design to finalize the protocol of FearLess, a psychological intervention targeting fear of cancer recurrence in primary malignant brain tumor patients and caregivers. Eligible participants (N=112) will be randomized to either: 1) immediate intervention or 2) delayed treatment control. Assessments will take place at baseline, Week 12, and Week 26.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Self-report a diagnosis of a primary malignant brain tumor (grade II-IV)
* >2 weeks post-cranial resection or biopsy
* Elevated Fear of Recurrence Distress Rating
* Primarily English speaking
* >/= 18 years of age at the time of enrollment

Caregivers:

* nonprofessional caregiver to a patient with a primary malignant brain tumor (grade II-IV)
* Elevated Fear of Recurrence Distress Rating
* Primarily English speaking
* >/= 18 years of age at the time of enrollment

Exclusion Criteria:

Patient / Caregiver Exclusion:

* Cognitive impairment that might prohibit active intervention engagement
* Inability to understand and provide informed consent
* Inability to attend virtual sessions due to unstable or no internet connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Study Enrollment | From screening to randomization allocation
  Feasibility of study enrollment using a multimodal recruitment approach will be assessed by comparing observed rates of screening completion, trial eligibility, trial enrollment (i.e., informed consent), and randomization allocation to pre-specified benchmarks.
Feasibility - Study Retention at 12 Weeks | From baseline assessment to 12 weeks
  Study retention will be measured by comparing observed rates of 12-week assessment completion to pre-specified benchmarks.
Feasibility - Study Retention at 24 Weeks | From baseline assessment to 24 weeks
  Study retention will be measured by comparing observed rates of 24-week assessment completion to pre-specified benchmarks.
Feasibility - Sustained Eligibility (Delayed Treatment Control Arm Only) | From baseline to 12-week assessment
  Feasibility of sustained trial eligibility will be assessed in the delayed treatment control arm only by comparing the proportion of participants who remain eligible at 12 weeks to a pre-determined threshold.
Acceptability - Intervention | From baseline to 12-week assessment in the Immediate Intervention arm; from 12-week assessment to 24-week assessment in the Delayed Treatment Control arm
  The acceptability of the intervention will be measured by comparing rates of intervention completion to pre-determined thresholds.
Acceptability - Intervention | From baseline to 12-week assessment in the Immediate Intervention arm; from 12-week assessment to 24-week assessment in the Delayed Treatment Control arm
  The acceptability of the intervention will be measured by comparing participant Acceptability Intervention Measure (AIM) scores to pre-determined thresholds. The AIM is a 4-item questionnaire that measures participant perception that a given treatment is agreeable, palatable, or satisfactory. Items are rated on a Likert scale from 1=Completely Agree to 5=Completely Disagree.
Acceptability - Trial Procedures | Week 24
  The acceptability of the trial procedures will be measured by comparing rates of participant satisfaction with randomization methodology and assessment procedures to pre-determined thresholds. The satisfaction measure consists of 4 Likert-scale items and 2 Yes/No items encompassing perceptions of satisfaction regarding randomization, intervention schedule, questionnaire burden, and honorarium.
Appropriateness - Interventionist Report | At 12-week assessment in the Immediate Intervention arm; at 24-week assessment in the Delayed Treatment Control arm
  Intervention appropriateness will be assessed by the study interventionists for each participant using the Intervention Appropriateness Measure (IAM). The IAM will be completed following each session; average score will be used for outcome analyses. The IAM is a 4-item standardized scale that measures the perceived fit, relevance, or compatibility of the intervention for a given practice setting, provider, or consumer, and/or perceived fit of the intervention to address a particular issue or problem. Items are rated on a Likert scale from 1=Completely Agree to 5=Completely Disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee R Loughan, Ph.D, Principal Investigator — Virginia Commonwealth University; Sarah E Braun, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No